CLINICAL TRIAL: NCT05546112
Title: Pilot Study to Explore the Efficacy and Safety of At-home Transcutaneous Electrical Nerve Stimulation in Insomnia
Brief Title: The Efficacy and Safety of At-home Transcutaneous Electrical Nerve Stimulation in Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ybrain Inc. (Industry)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YB-05
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Insomnia
Keywords: Transcutaneous electric nerve stimulation, TENS; Insomnia; Trigeminal nerve stimulation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Transcutaneous trigeminal nerve stimulation applied using clinical trial medical device (YPS-401B) for 20 minutes every night before going to bed, 28 times for 4 weeks at 1 time / 1 day
  Interventions: Device: Transcutaneous Trigeminal Electrical Nerve Stimulation using YPS-401B
- Control group (Sham Comparator): Sham stimulation applied using clinical trial medical device (YPS-401B) for 20 minutes every night before going to bed, 28 times for 4 weeks at 1 time / 1 day
  Interventions: Device: Sham Stimulation using YPS-401B

INTERVENTIONS:
Device: Transcutaneous Trigeminal Electrical Nerve Stimulation using YPS-401B — A device that improves insomnia symptoms by transcutaneously applying electrical stimulation including a pulse (10 kHz) burst waveform (10 Hz) to the forehead area to the trigeminal nerve
  Arms: Experimental group
Device: Sham Stimulation using YPS-401B — A device that is attached in the same way as a real medical device, but actually applies a shum stimulus
  Arms: Control group

SUMMARY:
The purpose of this study is to explore the effects and safety of transcutaneous electrical nerve stimulation (TENS) at home for patients diagnosed with insomnia on the improvement of insomnia and nervous stability.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 19 and under 65
* Those who meet the criteria for the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) for Insomnia
* Those with a score of 8 or higher based on the Korean version Insomnia severity index (ISI-K)
* A person whose sleeping environment and habits are regular, usually between 9:00 p.m. and 1:00 a.m., go to bed, lie down for 7 to 10 hours, and wake up between 5 and 10 a.m.
* In the case of patients who regularly take drugs for improving insomnia at least once a week, those who agree to discontinue taking the prohibited drugs in this study for a total of 5 weeks, 1 week to remove the drug effect after screening and 4 weeks for the clinical study period
* Persons who do not have a reason to prohibit the use of electrotherapy that can significantly affect biomarkers in relation to this study
* A person who voluntarily decides to participate and agrees in writing to abide by the precautions after hearing and understanding a sufficient explanation about this clinical trial

Exclusion Criteria:

* Those who have been diagnosed with sleep arousal disorders other than insomnia (hypersomnia disorder, narcolepsy, breathing-related sleep disorder, circadian rhythm sleep arousal disorder, parasomnia)
* Those who have insomnia due to physical illness or medications being taken
* Patients with major medical and neuropsychiatric diseases other than sleep disorders
* Persons who have had or are currently undergoing dental treatment with a history of implanting metallic materials into the upper body, such as the transcranial or face, neck, etc., where non-invasive electrical stimulation is difficult or impossible
* Compliance was evaluated by writing a sleep diary for 1 week from the start of treatment, and if a sleep diary of 3 days or less was kept for 1 week, it was excluded from the study.
* Those who have changed the type and dose of drugs used within the last 3 months, or the type and time of cognitive behavioral therapy
* If you are currently registered in another clinical trial or use another clinical trial drug or device within 60 days from the time of screening

Exclusion criteria prior to intervention (After the sleep diary for one week after the screening test, if the following criteria are met, the patient will be excluded from participation in the study before the intervention.)

* Those with less than 8 points based on the Korean version of Insomnia severity index (ISI-K)
* When writing a sleep diary for a week, if it is written for less than 3 days or has an irregular sleep schedule

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-04 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Insomnia Severity Index (ISI) | after 4 weeks
  Changes in Insomnia Severity Index (ISI) after 4 weeks from pretreatment:

SECONDARY OUTCOMES:
Remission rate of ISI | after 4 weeks
  Remission rate of ISI after 4 weeks compared to before treatment (Remission: ISI score of 7 or less)
Response rate of ISI | after 4 weeks
  Response rate of ISI after 4 weeks compared to before treatment (Response: ISI change of more than 7 points or 50% or more decrease)
Changes in Pittsburgh Slepp Quality Index (PSQI) | after 4 weeks
  Changes in Pittsburgh Slepp Quality Index (PSQI) after 4 weeks compared to before treatment
Changes in index of slepp diary | after 4 weeks
  Changes in index of sleep diary (sleep latency, bedtime, sleep time) after 4 weeks compared to before treatment
Changes in EEG index | after 4 weeks
  Changes in EEG index (absolute power, relative power) after 4 weeks compared to before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Changho Yoon, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: Undecided